CLINICAL TRIAL: NCT02862067
Title: SGLT2 Inhibition in Diabetic Patients With Heart Failure With Reduced Ejection Fraction
Brief Title: SGLT2 Inhibition in Diabetes and Heart Failure
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Other Study IDs: HM20007722; 16MCPRP31100003 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2016-08-01; First posted 2016-08-10 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Diabetes Mellitus, Type 2; Heart Failure, Systolic
Keywords: SGLT2; type 2 diabetes mellitus; systolic heart failure; heart failure with reduced ejection fraction
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Failure, Systolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Assessment of cardiorespiratory fitness — Assessment of cardiorespiratory fitness

SUMMARY:
To determine the effects of SGLT2 inhibition with empagliflozin on cardio-respiratory fitness in patients with systolic heart failure.

DETAILED DESCRIPTION:
The investigators hypothesize that Sodium-GLucose coTransporters (SGLT)-2 inhibition will improve cardio-respiratory fitness (CRF) in patients with systolic heart failure.

Participants treated with SGLT2 inhibitor Empagliflozin as standard of care will undergo assessments described below.

The investigators will measure CRF with a validated cardiopulmonary exercise test at baseline and after 4 weeks of treatment received as standard of care, to determine whether SGLT2 inhibition improves cardio-respiratory fitness assessed by changes in peak oxygen consumption (VO2)(mL/kg/min) and minute ventilation (VE)/carbon dioxide production (VCO2) slope, powerful independent clinical predictors of mortality in HF.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed clinical diagnosis of stable HF (NYHA class II-III) on maximally tolerated HF medical regimen including angiotensin-inhibitors, beta-adrenergic blockers, and loop diuretics
* Reduced left ventricular systolic function (LVEF<50%) documented in the prior 12 months
* Poorly controlled T2DM (HbA1c levels between 6.5% and 10.0%)
* 18 years old and older.

Exclusion Criteria:

* Type I diabetes;
* Type II diabetes with episodes of severe hypoglycemia <50 mg/dl by history, frequent changes in anti-diabetic regimen class in the past 3 months or with a prior episode of diabetic ketoacidosis (any time);
* Open label treatment with SGLT2 inhibitors (within the past month);
* Treatment with thiazolidinedione (within the past month), which may induce volume and sodium retention;
* Chronic Kidney Disease (GFR<45 ml/kg*min);
* Uncontrolled thyroid dysfunction (TSH<0.4>4.5 mcIU/ml);
* Pregnancy or of child-bearing potential;
* Active or recent (within 2 weeks) genital/urinal infection;
* Concomitant conditions or treatment which would affect completion or interpretation of the study including physical inability to walk or run on a treadmill such as decompensated HF (edema, NYHA class IV), significant ischemic heart disease, angina, arterial hypotension (BP systolic <90 mmHg), orthostatic arterial hypotension, arterial hypertension (resting BP systolic >160 mmHg), atrial fibrillation with rapid ventricular response, severe valvular disease, severe chronic obstructive or restrictive pulmonary disease, moderate- severe anemia (Hgb<10 g/dl);
* Abnormal BP or heart rate response, angina or ECG changes (ischemia or arrhy- thmias) occurring during baseline cardio-pulmonary exercise testing;
* Chronic use of oral corticosteroids;
* Inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 Diabetes Mellitus and Heart Failure with reduced Ejection Fraction or Systolic Heart Failure.
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2016-07; Primary Completion 2018-01-16 (Actual); Study Completion 2018-01-16 (Actual)

PRIMARY OUTCOMES:
SGLT2 inhibition effects on cardiorespiratory fitness (CRF). | 4 weeks
  To measure the effects of Empagliflozin on cardiorespiratory fitness in patients with type 2 diabetes and heart failure with reduced ejection fraction or systolic heart failure. The effects on CRF are determined by measuring changes in peak VO2 (mL/kg/min) and the VE/VCO2 slope.

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Carbone, PhD, MS, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
The investigators plan to present the data promptly upon analysis as an abstract to a national meeting and/or a manuscript.

REFERENCES:
- [Result] Carbone S, Canada JM, Billingsley HE, Kadariya D, Dixon DL, Trankle CR, Buckley LF, Markley R, Vo C, Medina de Chazal H, Christopher S, Buzzetti R, Van Tassell BW, Abbate A. Effects of empagliflozin on cardiorespiratory fitness and significant interaction of loop diuretics. Diabetes Obes Metab. 2018 Aug;20(8):2014-2018. doi: 10.1111/dom.13309. Epub 2018 Apr 23. PMID 29603546